CLINICAL TRIAL: NCT05764109
Title: AdhereNce to Cied Implantation GuidELInes: Cardiac rehAbilitation as a Window on Time-dependent Indications: an Observational Prospective Study (ANGELICA).
Brief Title: Adherence to Cied Implantation Guidelines and Cardiac Rehabilitation
Acronym: ANGELICA
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: CE 2296
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Left Ventricular Systolic Dysfunction; Myocardial Infarction
MeSH Terms: conditions — Ventricular Dysfunction, Left; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are limited data on how the guideline indications for ICD implantation are applied in clinical practice across Europe. Moreover, the impact of "time-dependence" of some indications to implantation on the guidelines adherence is still unknown.

Objective of the present observational study is the evaluation of the adherence to the scientific guidelines in patients with a time-dependent indication to ICD/CRT-D implantation admitted to an in-hospital cardiac rehabilitation program.

DETAILED DESCRIPTION:
Current guidelines recommend ICD implantation in patients at high risk of sudden cardiac death with either ischemic or non-ischemic heart disease. However, implantation rate of cardiac implantable electrical devices (CIED), especially ICD, CRT and CRT-D, is lower than expected and do not reflect guideline indications.

Several factors may justify the differences in ICD implantation rates across Europe and the gap between daily clinical practice and guidelines: economic restrictions, poor guidelines awareness, especially among referring cardiologists and general practitioners, and different guidelines adherence. The impact of "time-dependence" of some indications to CIED implantation on the guidelines adherence is still unknown.

Objective of the present observational study will be the evaluation of the adherence to the scientific guidelines in patients with a time-dependent indication to ICD/CRT-D implantation admitted to an in-hospital cardiac rehabilitation program.

This is a prospective, multicenter, observational study performed in 6 cardiac rehabilitation facilities.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an in-hospital cardiac rehabilitation program because of a recent index event;
* Provision of signed and dated informed consent form;
* Age ≥ 18 years.
* NYHA II-III class at the admittance in the cardiac rehabilitation facility;
* LVEF ≤ 40% at echocardiography at the admittance in the cardiac rehabilitation facility;
* Presence of a time-dependent indication to an ICD/CRT-D implantation:
* <3 month of optimal medical therapy;
* <40 days from the index myocardial infarction in patients with acute coronary syndrome;
* 3 months from the revascularization procedure in patients with surgery;
* <3 months in patients with a de-novo heart failure episode of no ischemic etiology.
* Patients who have already received an ICD/CRT-D for primary prevention before the admittance in the cardiac rehabilitation facility, despite a time-dependent indication to an ICD/CRT-D implantation;
* Indication to ICD-CRT-D implantation for primary prevention.

Exclusion Criteria:

* Inability to give informed consent (diminished understanding or comprehension);
* Age < 18 years;
* NYHA Class I or IV during the cardiac rehabilitation in-hospital stay;
* LVEF > 40% at echocardiography performed at the admittance in the cardiac rehabilitation facility
* Absence of a time-dependent indication to an ICD/CRT-D implantation;
* Indication to ICD-CRT-D implantation for secondary prevention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be those with LVEF <40% of both ischemic and non-ischemic etiology, NYHA class II-III, who, at the discharge from the hospital, do not show as satisfied the temporal windows suggested by the guidelines as useful for a conclusive LVEF evaluation:
  <3 month of optimal medical therapy; <40 days from the index myocardial infarction in patients with acute coronary syndrome; 3 months from the revascularization procedure in patients with surgery; <3 months in patients with a de-novo heart failure episode of no ischemic etiology.
Sampling Method: Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Rate of LVEF assessment | 3 months
  The evaluation of the rate of patients who will perform an echocardiography for LVEF assessment at the end of the time-window as suggested by the guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No